CLINICAL TRIAL: NCT01421667
Title: A Phase 2 Study of Brentuximab Vedotin in Relapsed or Refractory Non-Hodgkin Lymphoma (NHL)
Brief Title: A Study of Brentuximab Vedotin in Relapsed or Refractory Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGN35-012
Record Dates: First submitted 2011-08-19; First posted 2011-08-23 (Estimated); Results first posted 2016-10-13 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2015-06

CONDITIONS: Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, T-Cell
Keywords: Lymphoma, Large B-Cell, Diffuse; Antigens, CD30; Antibody-Drug Conjugate; Antibodies, Monoclonal; Lymphoma, Non-Hodgkin; Monomethyl auristatin E; Drug Therapy; Immunotherapy; Hematologic Diseases; Lymphoma; Lymphoma, B-Cell; Lymphoma, T-Cell
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, T-Cell; Hematologic Diseases; Lymphoma | interventions — Brentuximab Vedotin; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brentuximab vedotin+rituximab (Experimental)
  Interventions: Drug: brentuximab vedotin; Drug: rituximab
- Brentuximab vedotin (Experimental)
  Interventions: Drug: brentuximab vedotin

INTERVENTIONS:
Drug: brentuximab vedotin — 1.8 mg/kg every 3 weeks by IV infusion
  Other Names: Adcetris; SGN-35
Drug: rituximab — 375 mg/m2 every 3 weeks by IV infusion
  Arms: Brentuximab vedotin+rituximab

SUMMARY:
This is an open-label, multicenter, phase 2 clinical trial to evaluate the efficacy and safety of brentuximab vedotin as a single agent in patients with CD30-positive non-Hodgkin lymphoma (NHL) (Part A). The study will also evaluate the safety and efficacy of brentuximab vedotin in combination with rituximab in patients with relapsed or refractory diffuse large B-cell lymphoma (DLBCL) (Part B) as well as further evaluate correlation of CD30 expression and response in DLBCL (Part C).

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed NHL (DLBCL only for Parts B and C)
* Relapsed or refractory disease following at least 1 prior systemic therapy
* Measurable disease of at least 1.5 cm as documented by CT
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2

Exclusion Criteria:

* History of another primary invasive malignancy that has not been in remission for at least 3 years
* Current diagnosis of systemic or cutaneous anaplastic large cell lymphoma or mycosis fungoides
* B cell lymphoma previously treated with only single-agent rituximab (for patients receiving brentuximab vedotin only) or corticosteroids as monotherapy
* Known cerebral/meningeal disease

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2011-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corinna Palanca-Wessels, MD, PhD, Study Director — Seagen Inc.
Locations (34):
- United States (33):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope, Duarte, California
  - PMK Medical Group Inc., DBA Ventura County Hematology Oncology Specialists, Oxnard, California
  - Stanford Cancer Center, Stanford, California
  - Rocky Mountain Cancer Centers - Aurora, Aurora, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Cancer Specialists of North Florida - St. Augustine, Saint Augustine, Florida
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Minnesota Oncology Hematology P.A., Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - New York Oncology Hematology, P.C., Albany, New York
  - NYU Clinical Cancer Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic, The, Cleveland, Ohio
  - Willamette Valley Cancer and Research / USOR, Eugene, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - St. Francis Hospital, Greenville, South Carolina
  - Texas Oncology - Medical City Dallas, Dallas, Texas
  - Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology-Southwest Fort Worth, Fort Worth, Texas
  - MD Anderson Cancer Center / University of Texas, Houston, Texas
  - Texas Oncology - Seton Williamson, Round Rock, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Swedish Cancer Institute Medical Oncology, Edmonds, Washington
  - Seattle Cancer Care Alliance / University of Washington Medical Center, Seattle, Washington
  - Northwest Cancer Specialists, P.C., Vancouver, Washington
- British Columbia Cancer Agency - Vancouver Centre, Vancouver, British Columbia, Canada

REFERENCES:
- [Result] Horwitz SM, Advani RH, Bartlett NL, Jacobsen ED, Sharman JP, O'Connor OA, Siddiqi T, Kennedy DA, Oki Y. Objective responses in relapsed T-cell lymphomas with single-agent brentuximab vedotin. Blood. 2014 May 15;123(20):3095-100. doi: 10.1182/blood-2013-12-542142. Epub 2014 Mar 20. PMID 24652992
- [Result] Jacobsen ED, Sharman JP, Oki Y, Advani RH, Winter JN, Bello CM, Spitzer G, Palanca-Wessels MC, Kennedy DA, Levine P, Yang J, Bartlett NL. Brentuximab vedotin demonstrates objective responses in a phase 2 study of relapsed/refractory DLBCL with variable CD30 expression. Blood. 2015 Feb 26;125(9):1394-402. doi: 10.1182/blood-2014-09-598763. Epub 2015 Jan 8. PMID 25573987
- [Derived] Bartlett NL, Smith MR, Siddiqi T, Advani RH, O'Connor OA, Sharman JP, Feldman T, Savage KJ, Shustov AR, Diefenbach CS, Oki Y, Palanca-Wessels MC, Uttarwar M, Li M, Yang J, Jacobsen ED. Brentuximab vedotin activity in diffuse large B-cell lymphoma with CD30 undetectable by visual assessment of conventional immunohistochemistry. Leuk Lymphoma. 2017 Jul;58(7):1607-1616. doi: 10.1080/10428194.2016.1256481. Epub 2016 Nov 20. PMID 27868471

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Aug 2011 - Jun 2015
Pre-assignment Details: Four additional patients enrolled, but withdrew prior to receiving treatment.
Groups:
- CD30+ T-Cell NHL, BV: Part A - Brentuximab vedotin (BV) 1.8 mg/kg every 3 weeks by intravenous (IV) infusion in patients in with CD30-positive mature T-cell non-Hodgkin lymphomas (NHL)
- CD30+ B-Cell NHL, BV: Part A - Brentuximab vedotin (BV) 1.8 mg/kg every 3 weeks by intravenous (IV) infusion in patients with CD30-positive B-cell non-Hodgkin lymphomas (NHL), including CD30-positive diffuse large B-cell lymphoma (DLBCL) and other CD30-positive B-cell NHLs
- CD30u DLBCL, BV: Part C - Brentuximab vedotin (BV) 1.8 mg/kg every 3 weeks by intravenous (IV) infusion in patients with diffuse large B-cell lymphoma (DLBCL) with undetectable CD30 (CD30u)
- CD30+ DLBCL, BV+R: Part B - Brentuximab vedotin (BV) 1.8 mg/kg plus rituximab (R; first 8 cycles only) (375 mg/m2) every 3 weeks by intravenous (IV) infusion in patients with CD30-positive diffuse large B-cell lymphoma (DLBCL)
Period: Overall Study
Arm/Group | CD30+ T-Cell NHL, BV | CD30+ B-Cell NHL, BV | CD30u DLBCL, BV | CD30+ DLBCL, BV+R
Started | 35 | 68 | 53 | 16
Completed | 35 (Completed per protocol due to death [24] or study termination by sponsor [11]) | 66 (Completed per protocol due to death [45] or study termination by sponsor [21]) | 51 (Completed per protocol due to death [33] or study termination by sponsor [18]) | 15 (Completed per protocol due to death [7] or study termination by sponsor [8])
Not Completed | 0 | 2 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | CD30+ T-Cell NHL, BV | CD30+ B-Cell NHL, BV | CD30u DLBCL, BV | CD30+ DLBCL, BV+R | Total
Number analyzed (Participants) | 35 | 68 | 53 | 16 | 172
Age, Continuous [Median (Full Range); unit: years] | 64 [33 to 83] | 57 [16 to 85] | 65 [21 to 91] | 62 [22 to 78] | 63 [16 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 29 | 27 | 4 | 68
  Male | 27 | 39 | 26 | 12 | 104
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 7 | 1 | 14
  Not Hispanic or Latino | 32 | 65 | 46 | 15 | 158
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 0 | 2
  Asian | 1 | 3 | 4 | 0 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 5 | 6 | 4 | 0 | 15
  White | 29 | 55 | 41 | 15 | 140
  More than one race | 0 | 3 | 2 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Pathological Diagnosis [Number; unit: participants]
  Diffuse Large B-Cell Lymphoma (DLBCL) | 0 | 43 | 53 | 16 | 112
  Epstein-Barr Virus-Associated DLBCL of Elderly | 0 | 5 | 0 | 0 | 5
  Follicular Lymphoma | 0 | 3 | 0 | 0 | 3
  Gray Zone Lymphoma | 0 | 6 | 0 | 0 | 6
  Primary Mediastinal B-Cell Lymphoma | 0 | 6 | 0 | 0 | 6
  Post-Transplant Lymphoproliferative Disorder | 0 | 3 | 0 | 0 | 3
  Plasmablastic Lymphoma | 0 | 1 | 0 | 0 | 1
  T-Cell Rich B-Cell Lymphoma | 0 | 1 | 0 | 0 | 1
  Angioimmunoblastic T-cell Lymphoma | 13 | 0 | 0 | 0 | 13
  Peripheral T-Cell Lymphoma Not Otherwise Specified | 22 | 0 | 0 | 0 | 22
Transformed Disease from Prior Non-Hodgkin Lymphoma [Number; unit: participants]
  Yes | 1 | 14 | 11 | 5 | 31
  No | 34 | 54 | 42 | 11 | 141
Disease Stage [Number; unit: participants]
  Stage I | 2 | 4 | 1 | 1 | 8
  Stage II | 2 | 12 | 7 | 3 | 24
  Stage III | 13 | 17 | 11 | 6 | 47
  Stage IV | 14 | 31 | 33 | 6 | 84
  Unknown | 4 | 4 | 1 | 0 | 9
Bulky Disease (≥5 cm on at least one baseline index lesion) [Number; unit: participants]
  Yes | 5 | 27 | 35 | 4 | 71
  No | 30 | 41 | 18 | 12 | 101
Eastern Cooperative Oncology Group Performance Status (ECOG) [Number; unit: participants] — 0 = Normal activity; 1 = Symptoms but ambulatory; 2 = In bed <50% of the time; 3 = In bed >50% of the time; 4 = 100% bedridden; 5 = Dead
  participants
    0 | 7 | 25 | 10 | 9 | 51
    1 | 23 | 35 | 31 | 7 | 96
    2 | 5 | 7 | 12 | 0 | 24
    3-5 | 0 | 0 | 0 | 0 | 0
    Missing | 0 | 1 | 0 | 0 | 1
% CD30 Expression by Visual Immunohistochemistry (vIHC) [Median (Full Range); unit: percentage] — Percent CD30 expression by standard immunohistochemistry assessed visually by central laboratory (vIHC)
  percentage | 15 [0 to 95] | 35 [0 to 100] | 0 [0 to 10] | 50 [1 to 100] | 8 [0 to 100]
Refractory to Frontline Therapy [Number; unit: participants]
  Yes | 25 | 51 | 34 | 10 | 120
  No | 10 | 15 | 19 | 6 | 50
  Missing/Unknown | 0 | 2 | 0 | 0 | 2
Disease Status Relative to Most Recent Prior Therapy [Number; unit: participants]
  Refractory | 22 | 55 | 37 | 9 | 123
  Relapsed | 13 | 12 | 16 | 7 | 48
  Missing | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) by Investigator With Brentuximab Vedotin Monotherapy
Description: Percentage of participants treated with brentuximab vedotin monotherapy who achieved a best response of complete remission (CR, disappearance of all evidence of disease) or partial remission (PR, regression of greater than or equal to 50% of measurable disease and no new sites) per Cheson 2007 Revised Response Criteria for Malignant Lymphoma.
Time Frame: Up to approximately 3 years
Population: All participants who received treatment with brentuximab vedotin monotherapy and had both a baseline and at least one post-baseline disease assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- CD30+ T-Cell NHL, BV: Part A - CD30-positive T-cell non-Hodgkin lymphomas (NHL) include pathological diagnoses of angioimmunoblastic T-cell lymphoma (AITL) and peripheral T-cell lymphoma, not otherwise specified (PTCL-NOS).
- CD30+ Other B-Cell NHL, BV: Part A - CD30-positive other B-cell non-Hodgkin lymphomas (NHL) include pathological diagnoses of follicular lymphoma, gray zone lymphoma, primary mediastinal B-cell lymphoma (PMBL), post-transplant lymphoproliferative disease (PTLD), and plasmablastic lymphoma.
- CD30+ DLBCL, BV: Part A - CD30-positive diffuse large B-cell lymphoma (DLBCL) include pathological diagnoses of DLBCL, Epstein-Barr Virus (EBV)-associated DLBCL of the elderly, and T-cell rich B-cell lymphoma.
- CD30u DLBCL, BV: Part C - CD30u diffuse large B-cell lymphoma (DLBCL) includes only the pathological diagnosis of DLBCL.
Arm/Group | CD30+ T-Cell NHL, BV | CD30+ Other B-Cell NHL, BV | CD30+ DLBCL, BV | CD30u DLBCL, BV
Number analyzed (Participants) | 34 | 19 | 48 | 52
percentage of participants | 41 [24.6 to 59.3] | 26 [9.1 to 51.2] | 44 [29.5 to 58.8] | 31 [18.7 to 45.1]

2. Primary Outcome: Adverse Events by Severity, Seriousness, and Relationship to Treatment With Brentuximab Vedotin Plus Rituximab
Description: Counts of participants who had treatment-emergent adverse events (TEAE, defined as newly occurring or worsening after first dose on Study SGN35-012). Serious adverse events are reported from the time of informed consent. National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE version 4.03) were used to assess severity (1=mild, 2=moderate, 3=severe, 4=life-threatening/disabling, 5=fatal). Relatedness to study drug was assessed by the investigator (Yes/No). Participants with multiple occurrences of an adverse event within a category are counted once within the category.
Time Frame: Up to 3 years
Population: All participants who received treatment with brentuximab vedotin plus rituximab.
Measure: Number; unit: participants
Groups:
- CD30+ DLBCL, BV+R: Part B - CD30-positive diffuse large B-cell lymphoma (DLBCL) includes only the pathological diagnosis of DLBCL.
Arm/Group | CD30+ DLBCL, BV+R
Number analyzed (Participants) | 16
participants
  Any TEAE | 16
  TEAE Related to Study Drug | 15
  TEAE With Severity Grade >/=3 | 9
  Discontinued Treatment Due to Adverse Event | 2
  Serious Adverse Event | 3
  Serious Adverse Event Related to Study Drug | 3
  Deaths (Within 30 Days of Last Dose) | 1
  Chemistry Laboratory Abnormalities >/=Grade 3 | 1
  Hematology Laboratory Abnormalities >/=Grade 3 | 7

3. Secondary Outcome: Objective Response Rate (ORR) by Investigator With Brentuximab Vedotin Plus Rituximab
Description: Percentage of participants treated with brentuximab vedotin plus rituximab who achieved a best response of complete remission (CR, disappearance of all evidence of disease) or partial remission (PR, regression of greater than or equal to 50% of measurable disease and no new sites) per Cheson 2007 Revised Response Criteria for Malignant Lymphoma.
Time Frame: Up to approximately 3 years
Population: All participants who received treatment with brentuximab vedotin plus rituximab and had both a baseline and at least one post-baseline disease assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CD30+ DLBCL, BV+R
Number analyzed (Participants) | 12
percentage of participants | 50 [21.1 to 78.9]

4. Secondary Outcome: Complete Remission (CR) Rate by Investigator
Description: Percentage of participants treated with brentuximab vedotin monotherapy or brentuximab vedotin plus rituximab who achieved a best response of complete remission (CR, disappearance of all evidence of disease) per Cheson 2007 Revised Response Criteria for Malignant Lymphoma.
Time Frame: Up to approximately 3 years
Population: All participants who received brentuximab vedotin monotherapy or brentuximab vedotin plus rituximab and had both a baseline and at least one post-baseline disease assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CD30+ T-Cell NHL, BV | CD30+ Other B-Cell NHL, BV | CD30+ DLBCL, BV | CD30u DLBCL, BV | CD30+ DLBCL, BV+R
Number analyzed (Participants) | 34 | 19 | 48 | 52 | 12
percentage of participants | 24 [10.7 to 41.2] | 16 [3.4 to 39.6] | 19 [8.9 to 32.6] | 12 [4.4 to 23.4] | 17 [2.1 to 48.4]

5. Secondary Outcome: Duration of Objective Response With Brentuximab Vedotin Monotherapy by Kaplan-Meier Analysis
Description: Duration of complete remission (CR) or partial remission (PR), defined as time of initial response until disease progression or death. Response criteria per Cheson 2007 Revised Response Criteria for Malignant Lymphoma.
Time Frame: Up to approximately 3 years
Population: All participants who received treatment with brentuximab vedotin monotherapy and achieved a CR or PR.
Measure: Median (Full Range); unit: months
Arm/Group | CD30+ T-Cell NHL, BV | CD30+ Other B-Cell NHL, BV | CD30+ DLBCL, BV | CD30u DLBCL, BV
Number analyzed (Participants) | 14 | 5 | 21 | 16
months | 7.6 [1.3 to 36.1] | 1.6 [1.4 to 34] | 4.7 [0 to 22.7] | 4.7 [0.5 to 11.6]

6. Secondary Outcome: Duration of Complete Remission With Brentuximab Vedotin Monotherapy by Kaplan-Meier Analysis
Description: Duration of complete remission (CR), defined as time of initial response until disease progression or death. Response criteria per Cheson 2007 Revised Response Criteria for Malignant Lymphoma.
Time Frame: Up to approximately 3 years
Population: All participants who received treatment with brentuximab vedotin monotherapy and achieved CR
Measure: Median (Full Range); unit: months
Arm/Group | CD30+ T-Cell NHL, BV | CD30+ Other B-Cell NHL, BV | CD30+ DLBCL, BV | CD30u DLBCL, BV
Number analyzed (Participants) | 8 | 3 | 9 | 6
months | NA [1.8 to NA] — Not reached because too few events | 7.2 [1.6 to 34] | NA [2.2 to NA] — Not reached because too few events | 11.6 [1.4 to 11.6]

7. Secondary Outcome: Progression-Free Survival With Brentuximab Vedotin Monotherapy by Kaplan-Meier Analysis
Description: Progression-free survival, defined as time from start of study treatment to disease progression per investigator or death due to any cause
Time Frame: Up to approximately 3 years
Population: as for outcome 1
Measure: Median (Full Range); unit: months
Arm/Group | CD30+ T-Cell NHL, BV | CD30+ Other B-Cell NHL, BV | CD30+ DLBCL, BV | CD30u DLBCL, BV
Number analyzed (Participants) | 34 | 19 | 48 | 52
months | 2.5 [0.3 to 37.4] | 2.9 [0.6 to 36.3] | 4.0 [0.6 to 24.0] | 1.4 [0.4 to 15.6]

8. Secondary Outcome: Correlation Between Antitumor Activity of Brentuximab Vedotin Monotherapy and CD30 Expression
Description: Percentage of participants treated with brentuximab vedotin monotherapy who achieved a best response of complete remission (CR, disappearance of all evidence of disease), partial remission (PR, regression of greater than or equal to 50% of measurable disease and no new sites), or stable disease (SD, no new sites and no change in size of previous lesions) per Cheson 2007 Revised Response Criteria for Malignant Lymphoma. Patients are grouped by CD30-positivity or CD30u (undetectable CD30).
Time Frame: Up to 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CD30+ T-Cell NHL, BV | CD30+ Other B-Cell NHL, BV | CD30+ DLBCL, BV | CD30u DLBCL, BV
Number analyzed (Participants) | 34 | 19 | 48 | 52
percentage of participants
  Complete Remission (CR) | 24 [10.7 to 41.2] | 16 [3.4 to 39.6] | 19 [8.9 to 32.6] | 12 [4.4 to 23.4]
  Partial Remission (PR) | 18 [6.8 to 34.5] | 11 [1.3 to 33.1] | 25 [13.6 to 39.6] | 19 [9.6 to 32.5]
  Disease Control Rate (CR+PR+SD) | 59 [40.7 to 75.4] | 63 [38.4 to 83.7] | 69 [53.7 to 81.3] | 42 [28.7 to 56.8]

9. Secondary Outcome: Adverse Events by Severity, Seriousness, and Relationship to Treatment With Brentuximab Vedotin Monotherapy
Description: as for outcome 2
Time Frame: Up to 3 years
Population: All participants who received treatment with brentuximab vedotin monotherapy.
Measure: Number; unit: participants
Arm/Group | CD30+ T-Cell NHL, BV | CD30+ B-Cell NHL, BV | CD30u DLBCL, BV
Number analyzed (Participants) | 35 | 68 | 53
participants
  Any TEAE | 32 | 66 | 52
  TEAE Related to Study Drug | 28 | 62 | 39
  TEAE With Severity Grade >/=3 | 23 | 52 | 37
  Discontinued Treatment Due To Adverse Event | 6 | 7 | 4
  Serious Adverse Event | 15 | 34 | 22
  Serious Adverse Event Related to Study Drug | 5 | 15 | 7
  Deaths (Within 30 Days of Last Dose) | 3 | 5 | 6
  Chemistry Laboratory Abnormalities >/= Grade 3 | 8 | 16 | 10
  Hematology Laboratory Abnormalities >/= Grade 3 | 11 | 31 | 21

10. Secondary Outcome: Brentuximab Vedotin Antibody-Drug Conjugate (ADC) Concentration at End of Infusion (Ceoi) (Cycle 1)
Description: End of infusion concentration of ADC following the first dose of brentuximab vedotin
Time Frame: 1 day
Population: All patients who were treated with brentuximab vedotin monotherapy and had Ceoi of ADC results.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | CD30+ T-Cell NHL, BV | CD30+ B-Cell NHL, BV | CD30u DLBCL, BV
Number analyzed (Participants) | 32 | 63 | 50
ug/mL | 35.6 (25) | 40.0 (29) | 40.1 (43)

11. Secondary Outcome: Brentuximab Vedotin Antibody-Drug Conjugate (ADC) Trough Concentration (Ctrough) (Cycle 1)
Description: Trough concentration of ADC from 0 to 21 days following the first dose of brentuximab vedotin
Time Frame: 3 weeks
Population: All patients who were treated with brentuximab vedotin monotherapy and had Ctrough of ADC results.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | CD30+ T-Cell NHL, BV | CD30+ B-Cell NHL, BV | CD30u DLBCL, BV
Number analyzed (Participants) | 25 | 44 | 34
ug/mL | 0.44 (113) | 0.91 (119) | 0.86 (94)

12. Secondary Outcome: Maximum Concentration (Cmax) of Brentuximab Vedotin Monomethyl Auristatin E (MMAE) (Cycle 1)
Description: Maximum serum concentration of MMAE from 0 to 21 days following the first dose of brentuximab vedotin
Time Frame: 3 weeks
Population: All patients who were treated with brentuximab vedotin monotherapy and had Cmax of MMAE results.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | CD30+ T-Cell NHL, BV | CD30+ B-Cell NHL, BV | CD30u DLBCL, BV
Number analyzed (Participants) | 35 | 68 | 51
ng/mL | 4.71 (63) | 4.66 (88) | 3.95 (74)

13. Secondary Outcome: Time to Maximum Concentration (Tmax) of Brentuximab Vedotin Monomethyl Auristatin E (MMAE)
Description: Time of maximum serum concentration of MMAE from 0 to 21 days following the first dose of brentuximab vedotin
Time Frame: 3 weeks
Population: All patients who were treated with brentuximab vedotin monotherapy and had Tmax of MMAE results.
Measure: Median (Full Range); unit: days
Arm/Group | CD30+ T-Cell NHL, BV | CD30+ B-Cell NHL, BV | CD30u DLBCL, BV
Number analyzed (Participants) | 35 | 68 | 51
days | 1.90 [0.88 to 6.89] | 1.91 [0.91 to 20.90] | 1.94 [0.93 to 19.8]

14. Secondary Outcome: Baseline Soluble CD30 Expression
Description: Serum concentration of soluble CD30 before first dose of brentuximab vedotin
Time Frame: Baseline
Population: All patients who were treated with brentuximab vedotin monotherapy and had baseline sCD30 expression results.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | CD30+ T-Cell NHL, BV | CD30+ B-Cell NHL, BV | CD30u DLBCL, BV
Number analyzed (Participants) | 32 | 64 | 46
ng/mL | 1005.4 [89.4 to 26426.6] | 229.4 [33.2 to 21277.7] | 140.4 [53.4 to 1695.9]

ADVERSE EVENTS:
Time Frame: Up to 3 years
Description: TEAEs, defined as newly occurring (not present at baseline) or worsening after first dose of treatment
Groups:
- CD30+ NHL (T-Cell and B-Cell), BV: Brentuximab vedotin (BV) 1.8 mg/kg every 3 weeks by intravenous (IV) infusion in patients in with CD30-positive non-Hodgkin lymphomas (NHL), including T-cell lymphomas and B-cell lymphomas, as well as diffuse large B-cell lymphoma (DLBCL)
- CD30u DLBCL, BV: Brentuximab vedotin (BV) 1.8 mg/kg every 3 weeks by intravenous (IV) infusion in patients in Part C with diffuse large B-cell lymphoma (DLBCL) with undetectable CD30 (CD30u)
- CD30+ DLBCL, BV+R: Brentuximab vedotin (BV) 1.8 mg/kg plus rituximab (R; first 8 cycles only) (375 mg/m2) every 3 weeks by intravenous (IV) infusion in patients in Part B with diffuse large B-cell lymphoma (DLBCL)
Arm/Group | CD30+ NHL (T-Cell and B-Cell), BV | CD30u DLBCL, BV | CD30+ DLBCL, BV+R
Serious Adverse Events (participants affected / at risk) | 49/103 | 22/53 | 3/16
Other Adverse Events (participants affected / at risk) | 96/103 | 48/53 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CD30+ NHL (T-Cell and B-Cell), BV (N=103) | CD30u DLBCL, BV (N=53) | CD30+ DLBCL, BV+R (N=16)
Pneumonia (Infections and infestations) | 8 | 3 | 0
Sepsis (Infections and infestations) | 4 | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0
Breast cellulitis (Infections and infestations) | 0 | 1 | 0
Central nervous system abscess (Infections and infestations) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 1
Herpes zoster disseminated (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0
Mastoiditis (Infections and infestations) | 1 | 0 | 0
Meningoencephalitis herpetic (Infections and infestations) | 1 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Staphylococcal bacteremia (Infections and infestations) | 1 | 0 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 6 | 0
Angioimmunoblastic T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Peripheral T-cell lymphoma unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 3 | 0
Nausea (Gastrointestinal disorders) | 4 | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Jejunal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Pyrexia (General disorders) | 9 | 0 | 0
Asthenia (General disorders) | 0 | 2 | 0
Chest pain (General disorders) | 0 | 1 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypomagnasemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary alveolar hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 5 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 0
Brain mass (Nervous system disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 3 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Hallucination, visual (Psychiatric disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Lipase increased (Investigations) | 1 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Graft versus host disease (Immune system disorders) | 1 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CD30+ NHL (T-Cell and B-Cell), BV (N=103) | CD30u DLBCL, BV (N=53) | CD30+ DLBCL, BV+R (N=16)
Anemia (Blood and lymphatic system disorders) | 19 | 8 | 0
Neutropenia (Blood and lymphatic system disorders) | 31 | 13 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 5 | 1
Tachycardia (Cardiac disorders) | 5 | 3 | 1
Abdominal distension (Gastrointestinal disorders) | 6 | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 14 | 8 | 2
Constipation (Gastrointestinal disorders) | 19 | 15 | 2
Diarrhea (Gastrointestinal disorders) | 33 | 9 | 4
Nausea (Gastrointestinal disorders) | 28 | 17 | 8
Vomting (Gastrointestinal disorders) | 19 | 11 | 6
Asthenia (General disorders) | 10 | 3 | 1
Chills (General disorders) | 11 | 3 | 4
Fatigue (General disorders) | 43 | 17 | 4
Edema peripheral (General disorders) | 11 | 4 | 2
Pyrexia (General disorders) | 22 | 12 | 5
Upper respiratory tract infection (Infections and infestations) | 10 | 5 | 3
Urinary tract infection (Infections and infestations) | 2 | 7 | 0
Weight decreased (Investigations) | 12 | 6 | 0
Decreased appetite (Metabolism and nutrition disorders) | 23 | 9 | 0
Dehydration (Metabolism and nutrition disorders) | 7 | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 12 | 6 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 10 | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 5 | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 3 | 3
Dizziness (Nervous system disorders) | 6 | 5 | 2
Dysgeusia (Nervous system disorders) | 6 | 3 | 0
Headache (Nervous system disorders) | 13 | 6 | 3
Hypoesthesia (Nervous system disorders) | 7 | 2 | 1
Peripheral motor neuropathy (Nervous system disorders) | 7 | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 33 | 14 | 6
Anxiety (Psychiatric disorders) | 10 | 3 | 1
Insomnia (Psychiatric disorders) | 14 | 7 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 2 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 13 | 4 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 3 | 3
Night sweats (Skin and subcutaneous tissue disorders) | 8 | 8 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 5 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less